CLINICAL TRIAL: NCT06182410
Title: Defibrotide Prophylaxis of Transplant Associated-Thrombotic Microangiopathy in Patients With High-Risk Neuroblastoma Receiving Tandem Transplants
Brief Title: Defibrotide Prophylaxis of Transplant Associated-Thrombotic Microangiopathy for Neuroblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Industry sponsor decision
Sponsor: University of California, San Francisco (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 230822; NCI-2023-10277 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Transplant-Associated Thrombotic Microangiopathy; Neuroblastoma; High-risk Neuroblastoma; Thrombotic Microangiopathies
MeSH Terms: conditions — Neuroblastoma; Thrombotic Microangiopathies | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive Care (defibrotide) (Experimental): Participants receive defibrotide IV over 2 hours every six hours on days -8 to +21 during the first and second rounds of Hematopoietic stem-cell transplantation (HSCT).
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Given intravenously (IV)
  Other Names: Noravid

SUMMARY:
This phase II trial tests how well defibrotide works in preventing transplant-associated thrombotic microangiopathy (TA-TMA) in patients with high-risk neuroblastoma undergoing tandem transplants (hematopoietic stem cell transplant [HSCT]). TMA is a potential life-threatening complication of stem cell transplant. TMA is a possible side effect of the chemotherapy (conditioning regimen) patients receive to help treat high-risk neuroblastoma, because these medicines can sometimes damage the blood vessel walls in the body. This damage leads to formation of tiny blood clots in organs, especially the kidney. This then causes organ damage and leads to problems with how they function. This study may help researchers learn how defibrotide may help prevent TMA before it starts, or help treat it once it starts among patients with high-risk neuroblastoma undergoing tandem transplants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if administration of prophylactic defibrotide sodium (defibrotide) will prevent the development of TA-TMA in participants with high-risk neuroblastoma receiving tandem transplants compared to historic controls.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of defibrotide in the prevention of severe TA-TMA, as defined by any TA-TMA with one or more of the following complications:

Ia. Renal failure requiring dialysis; Ib. Pleural or pericardial effusion requiring any surgical intervention; Ic. Central nervous system dysfunction, including seizure, posterior reversible encephalopathy syndrome (PRES); Id. Pulmonary hypertension; Ie. Biopsy-proven gastrointestinal involvement with bleeding; If. Death not related to relapse of underlying neuroblastoma; II. To determine the incidence of grade ≥ 3 hemorrhage (per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0) in participants on prophylactic defibrotide (grade 3 hemorrhage = transfusion indicated; invasive intervention indicated; hospitalization).

EXPLORATORY OBJECTIVES:

I. To evaluate the incidence of hepatic sinusoidal obstructive syndrome (SOS) grade >= 2 (per Cairo criteria) with first and second HSCT.

II. To evaluate the percentage of patients who go on to second transplant compared to historic controls.

III. To evaluate median time in days to start of subsequent therapy (radiation and immunotherapy) and percent of patients who have delays compared to historic controls.

OUTLINE:

Participants receive defibrotide intravenously (IV) over 2 hours every 6 hours (Q6H) on days -8 to +21 during their first and second HSCT in the absence of unacceptable toxicity. After completion of study treatment, participants are followed until day +42 after second transplant and then every 2 weeks until 6 months after first HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1 - < 18 years old.
2. Participants must have high-risk neuroblastoma according to Children's Oncology Group (COG) risk classification at the time of initial diagnosis. Participants who were initially considered low or intermediate risk, but then reclassified as high risk are also eligible.
3. Participants may have had salvage therapies (i.e., meta-iodobenzylguanidine (MIBG), dinutuximab) after induction but cannot have progressive disease at start of 4.

   Planned tandem transplants with conditioning with cyclophosphamide-thiotepa and carboplatin-etoposide-melphalan on, or as per, NCT03126916 (ANBL1531) or other tandem-containing COG high-risk neuroblastoma trials.
4. Participants may be enrolled in upfront neuroblastoma protocol, but this is not required.
5. Upfront MIBG or other therapies is not a contraindication.
6. Organ function per institutional standard of care (SOC) guiding clearance for autologous HSCT.
7. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Life expectancy < 6 months.
2. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
3. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
4. Known bleeding diathesis or bleeding risk deemed by the treating physician to be a contraindication to administration of defibrotide or on concomitant therapeutic anticoagulation. Administration of heparin and/or alteplase for central line maintenance is allowed.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of transplant-associated thrombotic microangiopathy (TA-TMA) | Up to1 year
  The cumulative incidence of TA-TMA in participants will be compared to historical controls. The historic controls will be participants with high-risk neuroblastoma who underwent planned tandem transplant at University of California San Francisco (UCSF) between 2017 and 2023.

SECONDARY OUTCOMES:
Cumulative incidence of severe TA-TMA | Up to 1 year
  The cumulative incidence of severe TA-TMA in the patients enrolled on study compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Higham, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No